CLINICAL TRIAL: NCT00560105
Title: A Proof of Principal Randomized Controlled Eight-Week Study of the Safety and Efficacy of the Lung Flute in Adults With Chronic Obstructive Pulmonary Disease. A FDA 510(k) Equivalency Study
Brief Title: Randomized Controlled Eight-Week Study of the Safety and Efficacy of the Lung Flute
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Acoustics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1002
Record Dates: First submitted 2007-11-15; First posted 2007-11-19 (Estimated); Results first posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: COPD
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acapella (Active Comparator): The Active Comparator is the Acapella, a OPEP device
  Interventions: Device: Acapella
- Lung Flute (Experimental): The Active Comparator is the Lung Flute, a new indication of this device
  Interventions: Device: Lung Flute

INTERVENTIONS:
Device: Lung Flute — 8 weeks home use, twice daily
  Arms: Lung Flute
Device: Acapella — 8 weeks home use, twice daily
  Arms: Acapella

SUMMARY:
This is an eight-week, randomized, controlled, two arm parallel study. The study consists of, a screening visit, two weeks of intervention-free run-in randomization, clinic visits week 0, 1, 2, 4, 6, and 8 weeks during the intervention period to collect 24 hour sputum and to confirm techniques of device use and entries into daily diaries. Twenty-four (24) hour sputum samples will be collected and weighed at each clinic visit. In addition to clinic visits, subjects will be expected to make daily diary entries of COPD symptoms. Clinical evaluation will include adverse event surveillance, and St. Georges Respiratory questionnaire.

DETAILED DESCRIPTION:
No further details

ELIGIBILITY:
Inclusion Criteria:

* Age of over 40 with COPD

Exclusion Criteria:

* Children,
* New mothers; and
* Women intending to become pregnant

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Sethi, MD, Principal Investigator — VA Western NY Healthcare System
Locations (1):
- VA Western NY Healthcare System, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 45 subjects, of which 5 subjects either did not meet the initial inclusion/exclusion criteria (n=3) or did not meet the compliance criteria between the recruitment and randomization visit (n=2).
Pre-assignment Details: Of the 40 subjects who were randomized, 20 each were randomized to the 2 devices. Of these 40 subjects, 37 completed the study.
Groups:
- Acapella: Acapella : 8 weeks home use, twice daily The study consisted of a screening visit, two weeks of intervention-free run-in, a randomization visit and then on treatment clinic visits at 1, 2, 4, 6, and 8 weeks. Participants who met the inclusion/exclusion criteria on screening were enrolled and provided with a daily paper dairy to record symptoms and rescue albuterol use. In addition they were instructed to provide two 24 hr sputum collections over the next 2 weeks. A randomization visit was done within 2 weeks of the enrollment visit. Participants who were compliant with the 24 hr sputum collection and at least 50% of the daily dairy entries were randomized to either the Lung Flute® or the Acapella®
- Lung Flute: Lung Flute : 8 weeks home use, twice daily The study consisted of a screening visit, two weeks of intervention-free run-in, a randomization visit and then on treatment clinic visits at 1, 2, 4, 6, and 8 weeks. Participants who met the inclusion/exclusion criteria on screening were enrolled and provided with a daily paper dairy to record symptoms and rescue albuterol use. In addition they were instructed to provide two 24 hr sputum collections over the next 2 weeks. A randomization visit was done within 2 weeks of the enrollment visit. Participants who were compliant with the 24 hr sputum collection and at least 50% of the daily dairy entries were randomized to either the Lung Flute® or the Acapella®
Period: Overall Study
Arm/Group | Acapella | Lung Flute
Started | 20 | 20
Completed | 19 | 18
Not Completed | 1 | 2
Not completed — musculoskeletal chest discomfort with us | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acapella | Lung Flute | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (1.6) | 64.0 (2.4) | 62.5 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 15 | 13 | 28
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Safety and Efficacy of the Lung Flute Versus the Acapella for the Treatment of COPD in Adults. Twenty-four (24) Hour Dry Sputum Weight
Description: In order to test the overall treatment effect on dry sputum weight over the course of the study, mixed effects analysis were performed. These models allow us to account for the longitudinal nature of the data. We assumed that the observations collected within each patient were correlated; however, observations collected across patients were assumed to be independent. Dry sputum weights obtained prior to and at randomization were regarded as baseline measurements, while those obtained at week 1, 2, 4, 6 and 8 were examined for treatment effects.
Time Frame: 8 weeks
Population: All patient data included
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Acapella | Lung Flute
Number analyzed (Participants) | 19 | 18
g
  Sreening Event | 11.9 (2.8) | 14.5 (3.3)
  Week1 | 14.4 (3.1) | 14.3 (3.2)
  Week 2 | 14.5 (3.3) | 14.2 (3.2)
  Week 4 | 11.8 (2.8) | 15.2 (3.4)
  Week 6 | 11.7 (2.8) | 12.0 (2.8)
  Week 8 | 11.6 (2.7) | 12.1 (2.8)

2. Secondary Outcome: FEV1 - Baseline and Device Comparisons
Description: Spirometric data was collected primarily to document safety of the interventions. Pre- and Post-bronchodilator spirometry was obtained at the randomization visit and at Week 8.
Time Frame: 8 weeks
Population: A data collected included
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Acapella | Lung Flute
Number analyzed (Participants) | 19 | 18
liter
  Screening FEV1 | 1.43 (0.13) | 1.38 (0.14)
  Week 8 FEV1 | 1.49 (0.14) | 1.44 (0.19)

3. Secondary Outcome: Quality of Life Questionnaire/Daily Diary
Description: St. George's Respiratory Questionnaire (SGRQ) is a well validated, widely used health status questionnaire specific for COPD. Its minimum important difference (MID) is 4 units. Unit of measure: 0 to 100 (100 = more limitation)
Time Frame: 8 weeks
Population: All patient data included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acapella | Lung Flute
Number analyzed (Participants) | 19 | 18
units on a scale
  Screening | 45.5 (3.6) | 51.9 (3.1)
  Week 8 | 45.0 (4.2) | 47.2 (4.1)

4. Secondary Outcome: Change in CCQ Score
Description: The COPD Clinical Questionnaire (CCQ) is an objective validated tool to assess COPD symptoms. CCQ was measured at the randomization visit and at the end of the study visit at week 8. The CCQ is scaled 1 to 5. Five indicating no symptoms.
Time Frame: 8 weeks
Population: A patient population included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acapella | Lung Flute
Number analyzed (Participants) | 19 | 18
units on a scale
  Screening | 2.53 (0.20) | 3.24 (0.30)
  Week 8 | 2.29 (0.25) | 2.82 (0.26)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Acapella | Lung Flute
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No